CLINICAL TRIAL: NCT04158193
Title: Effectiveness of Acupuncture for Breast Cancer Related Lymphedema Patients: a Multicenter, Randomized, Sham-controlled Clinical Trial
Brief Title: Acupuncture for Breast Cancer Related Lymphedema
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tianjin University of Traditional Chinese Medicine (Other)
Collaborators: Baokang Hospital Affiliated to Tianjin University of Traditional Chinese Medicine (Unknown); Tianjin Medical University Cancer Institute and Hospital (Other); Gansu Provincial Cancer Hospital (Unknown); The Second Affiliated Hospital of Baotou Medical College (Other)
Responsible Party: Principal Investigator, Yi Guo, The Dean of Traditional Chinese medicine College, Tianjin University of Traditional Chinese Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2014CB543202-03
Record Dates: First submitted 2019-11-06; First posted 2019-11-08 (Actual); Last update posted 2019-11-08 (Actual); Status verified 2019-11

CONDITIONS: Breast Cancer Lymphedema
MeSH Terms: conditions — Breast Cancer Lymphedema | interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acupuncture group (Experimental): Subjects in the acupuncture group are given acupuncture treatment.
  Interventions: Other: acupuncture
- Sham acupuncture control group (Experimental): Subjects in the sham acupuncture control group are given non-acupoint shallow acupuncture.
  Interventions: Other: sham acupuncture

INTERVENTIONS:
Other: acupuncture — Subjects in acupuncture group will be received acupuncture treatment by inserting LI11, SJ5, SJ9, SJ13, SJ10, HT3, PC2, LI4, and LI15 on the affected limb and RN12, RN9, RN6, RN4, SP9, SP6. Needles will be remained for 30 minutes each time after DeQi sensation, one time a day，three times a week, the treatment will be lasted for 7 weeks.
  Arms: Acupuncture group
Other: sham acupuncture — Subjects in control group will be treated with non-acupoint shallow needling, points will be selected 1 cm at the radial direction from acupoint LI11, SJ5, SJ9, SJ13, SJ10, LI4, HT3, PC2, LI4, LI15; 2 cm at the left of acupoint RN12, RN9, RN6, RN4; 1 cm at the tibial direction from SP9, SP6.
  The needling manipulation is the same as that of the acupuncture group, but only the superficial skin of points are punctured. The depth of needling is less than 0.5 cm, and no manipulation will be performed after puncturing the skin. Needles will be remained for 30 minutes each time,one time a day，three times a week, the treatment will be lasted for 7 weeks.
  Arms: Sham acupuncture control group

SUMMARY:
The purpose of this study is to evaluate the clinical efficacy of acupuncture on chronic upper limb lymphedema in patients with breast cancer surgery

ELIGIBILITY:
Inclusion Criteria:

* At least 6 months after breast cancer surgery and presents with persistent breast cancer related upper extremity lymphedema for at least 3 months.
* Stage II lymphedema according to the 2016 consensus by the international society of lymphology.
* Women aged 18 to 80 years
* Out-patients
* Estimated life expectancy > 6 months
* Upper extremity lymphedema is defined a more than 10% volume difference between the affected and unaffected arms

Exclusion Criteria:

* Bilateral breast cancer related lymphedema
* Tumor metastasis or recurrent patient
* Patients who is undergoing chemotherapy, radiation therapy or targeted therapy
* Taking diuretic
* Upper extremity lymphedema reached more than 80% volume difference between the affected and unaffected arms
* History of primary lymphedema
* A diagnosis of severe heart, liver, kidney or hematologic disease
* Edema caused by upper extremity disability or other conditions such as heart failure, kidney disease or malnutrition
* Have hypoproteinemia
* Inflammation, scar, or trauma at the site of operation, or other active skin infections
* Unable to self-care, had a history of psychological disorders, or unable to communicate
* Received lymphedema treatment within the past 1 month
* Pregnancy or breastfeeding
* The presence of electronic medical device implants
* Deny to sign the informed written consent, or unwilling to conform to randomization
* Participation in other clinical trials during the study period

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-11 (Estimated); Primary Completion 2020-11 (Estimated); Study Completion 2021-04 (Estimated)

PRIMARY OUTCOMES:
Upper extremities volume | 7 weeks
  Volume measurement is also commonly used for the evaluation of lymphedema and the mean change in inter-limb volume difference from baseline to the end of the 7-week intervention will be included as primary outcome measure. The volume of the affected and unaffected limb will be measured by the volumetric measuring device (Baseline, America) using the water displacement method, which is considered as the most reliable method for volume measurements.

SECONDARY OUTCOMES:
Upper extremities circumferences | 7 weeks
  Various assessment methods are available but circumference measure is simple, convenient with low cost, and reliable. Therefore, the primary outcome measures will be the mean change in inter-limb circumference difference from baseline to the end of the 7-week intervention. The circumference will be measured by the measurement tape (Gulick Attachment, Baseline, America) at the wrist crease,5 cm above the wrist crease,10 cm above the wrist crease,15 cm above the wrist crease,20 cm above the wrist crease,25 cm above the wrist crease,30 cm above the wrist crease,35 cm above the wrist crease,where the lymphedema is most severe and its corresponding location on the unaffected limb.
VAS distension score | 7 weeks
  The VAS distension score is used to assess the degree of self-distension feeling at the affected upper extremities. It is evaluated by drawing a 10 cm horizontal line on the paper. One end of the horizontal line is 0, indicating no distension feeling; the other end is 10, indicating that the distension is unbearable; the middle part indicates different degrees of swelling. Let the subject draw a mark on the horizontal line according to the feeling of self-indicating degree of distension.
Common terminology criteria for adverse events (CTCAE 4.03) - edema limbs criteria | 7 weeks
  Common terminology criteria for adverse events (CTCAE 4.03) will be used to grade the severity of swelling using the edema limbs criteria. A grading of mild, moderate or severe swelling will be assessed based on the inter-limb circumference or volume discrepancy, anatomic architecture, appearance, or activities of daily living. The CTCAE 4.03 will allow us to evaluate the clinical significance of circumference change. Stages of lymphedema from the international society of lymphology Stages of lymphedema from the international society of lymphology will be used to grade the severity of lymphedema. Staging of 0, I, II, or III will be assessed based on severity of swelling, ability to reduce swelling by elevation, and skin changes.
The Disabilities of the Arm, Shoulder and Hand (DASH) Outcome Measure | 7 weeks
  Disabilities of the arm, shoulder, and hand (DASH) is a scale consists of two concepts: functional status (part A) andsymptoms (part B) respectively. The functional status part is further divided into three dimensions: physical, social, and psychological. The total score of the DASH ranges from 0 to 100 with higher scores representing worse symptoms and function. The DASH has good validity and responsiveness and it is recommended to assess upper extremity function in breast cancer survivors. The validated Chinese version of the DASH will be used in this study.
The MOS 36-Item Short-Form Health Survey (SF-36) | 7 weeks
  The medical outcome study 36-item short-form health survey (SF-36) is a commonly used instrument to assess quality of life that has good validity. The SF-36 includes the following eight concepts: physical functioning, role limitations due to physical problems, social functioning, bodily pain, general mental health, role limitations due to emotional problems, vitality, and general health perception. The validated Chinese version of the SF-36 will be used in this study.